CLINICAL TRIAL: NCT04161170
Title: Validation of Diabetes Management Effectiveness of Digital Integrated Healthcare Platform Utilizing AI-based Dietary Management Solution and Real-time Continuous Glucose Monitoring System
Brief Title: Digital Integrated Healthcare Platform in Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jae Hyeon Kim, MD, PhD, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-05-028-007
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes
Keywords: Continuous glucose monitoring system; Artificial intelligence; Diabetes; Digital healthcare; Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Control group A: no intervention Interventional group B: digital integrated healthcare platform Interventional group C: digital integrated healthcare platform + CGMS apply + medical team monitoring + educational intervation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control A (No Intervention): no intervention conventional diabetes treatment and clinic visit every 3 months
- Intervention B (Active Comparator): apply digital integrated healthcare platform clinic visit every 3 months
  Interventions: Device: Digital integrated healthcare platform
- Intervention C (Experimental): apply digital integrated healthcare platform, CGMS, and medical team monitoring, and education clinic visit every 3 months
  Interventions: Device: Digital integrated healthcare platform

INTERVENTIONS:
Device: Digital integrated healthcare platform — Digital Integrated Healthcare Platform Utilizing AI-based Dietary Management Solution and Real-time Continuous Glucose Monitoring system
  Arms: Intervention B; Intervention C

SUMMARY:
In this three multicenter clinical trial, investigators will study the efficacy of digital integrated healthcare platform and CGMS (continuous glucose monitoring system) on diabetes management in patients with Type 2 diabetes. The platform is based on monitoring and intervention by medical staff using AI (aritificial intelligence)-based diet management solution.

The study group includes 3 groups; a total of 294 participants with 1:1:1 randomized allocation: Control group A (no intervention and conventional diabetes management with regular outpatiant clinic visit every 3 months), Interventional group B (applying digital integrated healthcare platform by themselves, no monitoring and intervention by medical staff), and Interventional group C (applying digital integrated healthcare platform based on monitoring and intervention by medical staff using AI-based diet management solution and applying CGMS).

This parallel study will be conducted for 48 weeks.

DETAILED DESCRIPTION:
The reason why it is difficult to improve the lifestyle of patients with diabetes using existing digital healthcare applications (apps) is that there is a limit of sustainability that most people do not continue to use digital healthcare apps, thus, it can be possible only with monitoring and intervention by medical staff.

Not only users, but also medical staff can access integrated biometric data on the digital integrated healthcare platform so that individual patient-specific management systems that monitor and intervene can continuously motivate patients to manage themselves. Also, it could be a prerequisite for the successful management of patients with diabetes using digital healthcare apps, many existing apps have been identified as failure cases in previous studies. In this clinical trial, investigators will study the efficacy of digital integrated healthcare platform based on monitoring and intervention by medical staff using AI (aritifical intelligence)-based diet management solution.

In addition, in this clinical trial, the latest medical device, real-time continuous glucose monitoring system (CGMS) will be applied to monitor blood glucose levels. It has been reported that glucose level is well controlled when the number of self blood glucose measurement is performed frequently, but in practice, patients have time and space limitation in self blood glucose measurement, and it is difficult to change the management pattern of patients by encouraging self blood glucose measurement. Therefore, by applying a CGMS every three months, not only the patient but also the medical staff can access the 24-hour blood glucose values, and can actively participate in the blood sugar management of the patients. Therefore, investigators plan to conduct clinical trial using digital integrated healthcare platform using AI-based diet management solution and real-time CGMS

ELIGIBILITY:
Inclusion Criteria:

* 19~70 aged patients with type 2 diabetes
* Patients who have not taken diabetic medications for more than 4 weeks and patients who have taken at least one type of oral hypoglycemic agents at same dosage for more than 12 weeks
* Those who have glycated hemoglobin within 7.0% to 8.5% within the last 3 months
* overweight or obese: BMI (body mass index) ≥ 23 kg / m2
* Those who have agreed to use medical record and participate research by applying the digital integrated healthcare platform
* Those who voluntarily signed the consent form after listening the explanation of the clinical trial.

Exclusion Criteria:

* Diabetes other than type 2 diabetes, including type 1 diabetes and gestational diabetes
* Those who are receiving insulin or GLP-1 agonist other than oral hypoglycemic agents
* Uncontrolled chronic liver disease (hemochromatosis, liver cancer, autoimmune liver disease, cirrhosis of the liver, viral hepatitis-includes all A, B and C, Wilson's disease)
* Those with acute renal failure (up to 1.5 times higher than existing serum creatinine)
* Those with mental illness (schizophrenia, depression, bipolar disorder, etc.)
* Those who are currently taking weight loss agents
* Those who had alcohol or drug addiction within the last three months
* Those who are taking medications that may affect glucose metabolism (eg, corticosteroids, immunoreactive drugs, etc.)
* Those who are pregnant or lactating and planning to become pregnant during the clinical trial (women of childbearing age may agree to the contraceptive plan).
* Those who are deemed inappropriate for participation in clinical trials

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of HbA1c (glycated hemoglobin) at 6months from baseline | Change of HbA1c (glycated hemoglobin) at 6months from baseline
  Change of HbA1c (glycated hemoglobin) at 6months from baseline

SECONDARY OUTCOMES:
HbA1c | glycated hemoglobin at baseline, 3, 6, 12 months
  glycated hemoglobin
number of intervention for education in interventinal group C | number of intervention for education in interventinal group C at baseline, 3, 6, 12 months
  The number of educational intervention by digital integrated healthcare platform
hypoglycemic events | hypoglycemic events at baseline, 3, 6, 12 months
  the number of hypoglycemic events
adverse events | adverse events at baseline, 3, 6, 12 months
  the number and types of hypoglycemic events
patient satisfaction questionnaire score | patient satisfaction questionnaire score at baseline, 3, 6, 12 months
  patient satisfaction questionnaire score includes 8 questions and each question has score range 0 (min) - 6 (max). For questions number 2 and 3, higher score mean worse outcome in hypoglycemia but for the rest of questions, higher scores mean better outcome in diabetes management.
body weight | body weight at baseline, 3, 6, 12 months
  body weight
BMI (body mass index) | BMI at baseline, 3, 6, 12 months
  BMI (body mass index)
body fat (%) | body fat (%) at baseline, 3, 6, 12 months
  body fat (%)
step count | average step count at baseline, 3, 6, 12 months
  step count
burned calories | average burned calories at baseline, 3, 6, 12 months
  burned calories
walking distances | average walking distances at baseline, 3, 6, 12 months
  walking distances
intake calories | intake calories at baseline, 3, 6, 12 months
  intake calories
fasting glucose level | average fasting glucose level at baseline, 3, 6, 12 months
  fasting glucose level
total cholesterol level | total cholesterol level at baseline, 3, 6, 12 months
  total cholesterol level
HDL cholesterol level | HDL cholesterol level at baseline, 3, 6, 12 months
  HDL cholesterol level
Triglycerides level | Triglycerides level at baseline, 3, 6, 12 months
  Triglycerides level
LDL cholesterol level | LDL cholesterol level at baseline, 3, 6, 12 months
  LDL cholesterol level
mean glucose level by CGMS (continuous glucose monitoring system) in interventional group C | mean glucose level by CGMS at baseline, 3, 6, 12 months
  mean glucose level by CGMS in interventional group C
glycemic variability by CGMS in interventional group C | glycemic variability by CGMS at baseline, 3, 6, 12 months
  glycemic variability by CGMS in interventional group C
standard deviation by CGMS in interventional group C | standard deviation by CGMS at baseline, 3, 6, 12 months
  standard deviation by CGMS in interventional group C
average applying time of CGMS in interventional group C | average applying time of CGMS at baseline, 3, 6, 12 months
  average applying time of CGMS in interventional group C
time in range of <54mg/dL by CGMS in interventional group C | time in range of <54mg/dL by CGMS at baseline, 3, 6, 12 months
  time in range of <54mg/dL by CGMS in interventional group C
time in range of <70mg/dL by CGMS in interventional group C | time in range of <70mg/dL by CGMS at baseline, 3, 6, 12 months
  time in range of <70mg/dL by CGMS in interventional group C
time in range of 70-180 mg/dL by CGMS in interventional group C | time in range of 70-180 mg/dL by CGMS at baseline, 3, 6, 12 months
  time in range of 70-180 mg/dL by CGMS in interventional group C
time in range of >180 mg/dL by CGMS in interventional group C | time in range of >180 mg/dL by CGMS at baseline, 3, 6, 12 months
  time in range of >180 mg/dL by CGMS in interventional group C
time in range of >250 mg/dL by CGMS in interventional group C | time in range of >250 mg/dL by CGMS at baseline, 3, 6, 12 months
  time in range of >250 mg/dL by CGMS in interventional group C

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hyeon Kim, MD PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee YB, Kim G, Jun JE, Park H, Lee WJ, Hwang YC, Kim JH. An Integrated Digital Health Care Platform for Diabetes Management With AI-Based Dietary Management: 48-Week Results From a Randomized Controlled Trial. Diabetes Care. 2023 May 1;46(5):959-966. doi: 10.2337/dc22-1929. PMID 36821833
- [Derived] Park SW, Kim G, Hwang YC, Lee WJ, Park H, Kim JH. Validation of the effectiveness of a digital integrated healthcare platform utilizing an AI-based dietary management solution and a real-time continuous glucose monitoring system for diabetes management: a randomized controlled trial. BMC Med Inform Decis Mak. 2020 Jul 10;20(1):156. doi: 10.1186/s12911-020-01179-x. PMID 32650771